CLINICAL TRIAL: NCT05140616
Title: Study of Chidamide in the Treatment of Steroid-resistant/Steroid-dependent Severe cGVHD
Brief Title: Study of Chidamide for Steroid-resistant/Steroid-dependent Severe cGVHD
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: cGVHD-01
Record Dates: First submitted 2021-07-06; First posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-05

CONDITIONS: Safety and Efficacy
MeSH Terms: interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study of Chidamide in the Treatment of Steroid-resistant/Steroid-dependent Severe cGVHD (Experimental): Subjects receive twice a week dose of 15mg of Chidamide tablets
  Interventions: Drug: Chidamide

INTERVENTIONS:
Drug: Chidamide — After screening according to inclusion and exclusion criteria, patients meeting the criteria were enrolled. Treatment regimen: Chidamide 15mg biw po, lasted for 8 weeks. Pretransplant use of Chidamide for reasons other than cGVHD, such as for the treatment of leukemia or lymphoma, was permitted.All patients received systemic corticosteroid therapy for cGVHD prior to and during the study; concomitant use of other immunosuppressive therapies was also permitted, however, pre-existing corticosteroid and immunosuppressant doses must have been stable for 14 days before initiating Chidamide. Doses of concomitant corticosteroids and immunosuppressants could be tapered during the study as clinically indicated.

SUMMARY:
Allogeneic hematopoietic stem cell transplantation (Allo-HSCT) is one of the most important and effective methods for the treatment of hematologic malignancies.Chronic graft-versus-host disease (cGVHD) is a serious complication of allogeneic stem cell transplantation with few effective options available after failure of corticosteroids. It is a leading cause of late nonrelapse mortality for transplant patients, also contributing to morbidity and a decrease in quality of life.Corticosteroids, the standard frontline treatment, are typically administered for a median of 2 to 3 years, leading to substantial morbidity. An effort to decrease corticosteroid doses has led to their use in combination with other immunosuppressants, such as cyclosporine, tacrolimus, and sirolimus, in frontlineor second-line settings, despite a lack of clinical evidence supporting additional efficacy after combining these agents with corticosteroids. B and T cells play a rolein the pathophysiology of cGVHD. Previous studies have shown that low-dose histone deacetylase inhibitors (HDACi) have a negative immune regulation in GVHD while maintain the GVL effect. Chidamide is one of new HDACis in China, the previous studies suggested that low dose Chidamide could reduce condition of cGVHD mice by regulating the immune homeostasis of follicular helper T (Tfh) cells. Chidamide also has effects on the regulation of antigen presenting cells, the activation donor T cells, the release of proinflammatory cytokines and the function of Treg cells. Furthermore, low-dose Chidamide has the potential to maintain GVL effects. In preclinical models,Chidamide reduced severity of cGVHD. Based on the biological rationale and preclinical data, a study was designed to evaluate the safety and efficacy of Chidamide in patients with cGVHD who was steroid-resistant/steroid-dependent .

DETAILED DESCRIPTION:
Promoting graft-versus-leukemia (GVL) effect and inhibiting chronic graft-versus-host disease (cGVHD), is the key to improve the efficacy of allogeneic hematopoietic stem cell transplantation (allo-HSCT). Previous studies have shown that low-dose histone deacetylase inhibitors (HDACi) have a negative immune regulation in aGVHD while maintain the GVL effect. Chidamide is one of new HDACis in China, its immune regulatory role in cGVHD is unclear. The results suggested that low dose Chidamide could reduce condition of cGVHD mice by regulating the immune homeostasis of follicular helper T (Tfh) cells. Chidamide also has effects on the regulation of antigen presenting cells, the activation donor T cells, the release of proinflammatory cytokines and the function of Treg cells. Furthermore, low-dose Chidamide has the potential to maintain GVL effects.

On this basis,a study was designed to evaluate the safety and efficacy of Chidamide in patients with cGVHD who was steroid-resistant/steroid-dependent.To Evaluate the Safety and Tolerability of Chidamide in Steroid Dependent/Refractory cGVHD.Number of participants with dose-limiting toxicities as a measure of safety profile to determine recommended dose of Chidamide.

Inclusion Criteria:

1. The disease progressed after at least 1 week of treatment with ≥ 1 mg/kg/d prednisone based immunosuppressive therapy;
2. The disease did not improve after at least 1 month of immunosuppressive therapy with ≥ 1 mg·kg once every 2 days or ≥ 0.5 mg/kg/d prednisone;
3. Gocorticoid dependence: Prednisone with > 0.25 mg/kg/d or > 0.5 mg·kg every 2 days after at least 8 weeks of glucocorticoid-based immunosuppressant therapy is required to prevent recurrence or progression.
4. Patients with severe glucocorticoid-resistant/dependent cGVHD who have poor response to second-line treatment drugs (mycophoranate, high-dose glucocorticoid, extracorporeal light therapy, sirolimus, imatinib, azathiopurine, thalidomide, rituximab, anti-CD25, etc.).
5. Ages 18-59
6. ECOG score 0-3
7. Expected survival longer than 6 months
8. The patient who signed the informed consent must be able to understand and willing to participate in the study, and must sign the informed consent.

Exclusion Criteria:

1. Basic diseases of important organs: such as myocardial infarction, chronic cardiac insufficiency, decompensated liver insufficiency, renal insufficiency, etc.;Clinically uncontrolled active infections (including bacterial, fungal or viral infections), but not those under effective medication;
2. Malignant tumors with other progression;
3. Cardiac dysfunction patients: ejection fraction (EF) < 30%, NYHA standard, cardiac dysfunction grade Ⅲ or above;
4. Pregnant or lactating women;
5. People undergoing clinical trials of other drugs; After screening according to inclusion and exclusion criteria, patients meeting the criteria were enrolled. Treatment regimen: Chidamide 15mg biw po, lasted for 8 weeks. Pretransplant use of Chidamide for reasons other than cGVHD, such as for the treatment of leukemia or lymphoma, was permitted.All patients received systemic corticosteroid therapy for cGVHD prior to and during the study; concomitant use of other immunosuppressive therapies was also permitted, however, pre-existing corticosteroid and immunosuppressant doses must have been stable for 14 days before initiating Chidamide. Doses of concomitant corticosteroids and immunosuppressants could be tapered during the study as clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

1. The disease progressed after at least 1 week of treatment with ≥ 1 mg/kg/d prednisone based immunosuppressive therapy;
2. The disease did not improve after at least 1 month of immunosuppressive therapy with ≥ 1 mg·kg once every 2 days or ≥ 0.5 mg/kg/d prednisone;
3. Gocorticoid dependence: Prednisone with > 0.25 mg/kg/d or > 0.5 mg·kg every 2 days after at least 8 weeks of glucocorticoid-based immunosuppressant therapy is required to prevent recurrence or progression.
4. Patients with severe glucocorticoid-resistant/dependent cGVHD who have poor response to second-line treatment drugs (mycophoranate, high-dose glucocorticoid, extracorporeal light therapy, sirolimus, imatinib, azathiopurine, thalidomide, rituximab, anti-CD25, etc.).
5. Ages 18-59
6. ECOG score 0-3
7. Expected survival longer than 6 months
8. The patient who signed the informed consent must be able to understand and willing to participate in the study, and must sign the informed consent.

Exclusion Criteria:

1. Basic diseases of important organs: such as myocardial infarction, chronic cardiac insufficiency, decompensated liver insufficiency, renal insufficiency, etc.;Clinically uncontrolled active infections (including bacterial, fungal or viral infections), but not those under effective medication;
2. Malignant tumors with other progression;
3. Cardiac dysfunction patients: ejection fraction (EF) < 30%, NYHA standard, cardiac dysfunction grade Ⅲ or above;
4. Pregnant or lactating women;
5. People undergoing clinical trials of other drugs;

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-05-31 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
To Evaluate the Safety and Tolerability of Chidamide in Steroid Dependent/Refractory cGVHD.Number of participants with dose-limiting toxicities as a measure of safety profile to determine recommended dose of Chidamide. | up to 12 months
  The primary end point was safety, tolerability and efficacy,which included the number of dose limiting toxicities occurring on Chidamide. The primary efficacy endpoint was the best overall cGVHD response rate on 3 montns and 6 months, which was defined as the proportion of all patients who achieved a complete response (CR) or partial response (PR).
  It will begin with the evaluation of the safety of the dose (Chidamide 15mg biw po, lasted for 8 weeks) with the potential for subsequent dose reductions if dose limiting toxicities (DLTs) are detected. A dose limiting toxicity (DLT) is defined as any drug-related hematologic or non-hematologic toxicity Grade 3 or higher.
  Best overall cGVHD response rate is defined as the proportion of subjects who achieve a NIH-defined complete response (CR) or partial response (PR) during the study.

CONTACTS AND LOCATIONS:
Overall Officials: depei Wu, Study Chair — the first affiliated hospital of Soochow Uninersity
Locations (1):
- First Affiliated Hospital,Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No